CLINICAL TRIAL: NCT00431925
Title: Can Cytokines Predict the Severity of Acute Mucositis and the Need for PEG During Chemo-Radiation Treatment to Head and Neck Cancer?
Brief Title: Can Cytokines Predict the Severity of Acute Mucositis and the Need for Gastrostomy Tubes (PEG)?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: MucoCyt- HMO-CTIL
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-02

CONDITIONS: Oral Mucositis; Xerostomia; Weight Loss; Head and Neck Cancer
Keywords: head and neck cancer; radiation therapy; chemotherapy; mucositis; cytokines; gastrostomy; radiotherapy
MeSH Terms: conditions — Stomatitis; Xerostomia; Weight Loss; Head and Neck Neoplasms; Mucositis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Mucositis and xerostomia are the most common complications of head and neck (H&N) irradiation, and the combination of chemotherapy and radiation therapy is associated with a significantly higher rate of complications.

Mucositis usually develops during the second or third week of a course of standard radiotherapy, and the pain it causes peaks between the third and last week of treatment. The pain then persists for at least one month following the completion of therapy, and may be so overwhelming that it prevents patients from swallowing food and fluids. The patient is therefore at a risk to develop malnutrition, and must be treated vigorously. In this respect, the use of gastrostomy tubes (PEG) has been shown to be beneficial.

Completion of the full course of irradiation, without interruption, is important for achieving best possible results in cancer of the H&N. It is therefore essential to identify and refer patients at risk to receive effective and timely nutritional intervention.

Since mucositis represents a clinical continuum which differs between patients, it is difficult to assess before-hand which patients will be at risk.

There is no simple laboratory tool available, which could predict which patients are susceptible to develop severe mucositis and dysphagia, and eventually will require a feeding gastrostomy.

The first phase of mucositis, inflammation, results in the production of pro-inflammatory cytokines such as interleukin-1 (IL-1) and tumor necrosis factor-alpha (TNF-α).

In general, the inflammatory cytokines IL-1, interleukin-6 (IL-6) and TNF-α are elevated in inflammatory conditions and are found in increased levels in blood and tissue fluid during inflammation, while anti-inflammatory cytokines are produced in a decreased manner.

The main purpose of this study is to find the best indicators and prognosticators of mucositis occurring in the healthy oral tissues of H&N cancer patients receiving treatment, and to understand the cytokines balance mechanism of action.

Assuming there is a correlation between high cytokines levels during inflammation and the severity of radiation induced mucositis, finding these prognostic factors may help us predict during the first part of the treatment the need for PEG, placing it prior to the complications associated with severe mucositis on one hand, and avoiding unnecessary procedures on the other hand.

DETAILED DESCRIPTION:
Mucositis has a significant detrimental effect on patient's quality of life in terms of pain, ability to eat, to swallow and talk. It may be so severe that an interruption of therapy is required, consequently influencing tumor response and overall patient outcome.

The degree of mucositis varies between different patients: some patients may develop a limited condition, confined to patches of mildly sore erythematous mucosa, while others may experience diffuse areas of painful ulceration.

In the more severe cases, pain may be so overwhelming that it prevents patients from swallowing food and fluids. The patient is therefore at a risk to develop malnutrition, and must be treated vigorously. In this respect, the use of gastrostomy tubes (PEG) has been shown to be beneficial.

Another aspect of radiation induced mucositis is its health-care costs. Patients with more severe mucositis have statistically greater outpatient support costs; these include maintenance of appropriate nutritional and hydration support, such as placement of gastrostomy tubes. In the U.S, the mucositis overall medical costs are in the order of approximately $3000±$1000, per treatment.

Completion of the full course of irradiation, without interruption, is important for achieving best possible results in cancer of the H&N. It is therefore essential to identify and refer patients at risk to receive effective and timely nutritional intervention.

Since mucositis represents a clinical continuum which differs between patients, it is difficult to assess before-hand which patients will be at risk to develop severe mucositis during the course of radiotherapy. In today's practice, patients undergoing radiation therapy of the H&N will undergo feeding gastrostomy by the treating physician prior to the treatment if he will anticipate severe mucositis, based on the radiation fields, the chemotherapy used, and his prior experience. Some of these procedures were eventually unnecessary. In cases where gastrostomy was not placed a priory, the common practice is monitoring the patients during treatment. If their weight loss exceeds 10% of their initial body weight, a feeding gastrostomy is recommended (at this time point, the mucositis is usually severe, and many patients need admission for fluid administration and semi-urgent procedure).

Unfortunately, there is no simple laboratory tool available, which could predict which patients are susceptible to develop severe mucositis and dysphagia, and eventually will require a feeding gastrostomy.

Mucositis develops in four successive phases: an inflammation phase, an epithelial phase, an ulceration phase and lastly, a healing phase.

The first phase, inflammation, is also entitled "the initial tissue injury phase", and it results in the production of pro-inflammatory cytokines such as IL-1 and TNF-α .

In general, the inflammatory cytokines IL-1, IL-6 and TNF-α are elevated in inflammatory conditions and are found in increased levels in blood and tissue fluid during inflammation, while anti-inflammatory cytokines are produced in a decreased manner.

In breast cancer patients, it has been shown that changes in cytokines levels, Including IL-1β and IL-6, also correspond with the response of the malignant tissue to treatment. In this case, a good clinical response to therapy has been associated with decreases in IL-1β and IL-6 levels, versus increases in their levels which have been associated with the progression of the disease. Furthermore, tumor markers such as the cytokeratin TPS, have been shown to be sensitive in assessing the tumor's response to therapy and the patient's prognosis.

It should be emphasized though, that the findings cited above reflect the response of tumor cells to therapy, while the proposed project deals with radiation effects on both normal tissues and tumor.

The main purpose of this study is to find the best indicators and prognosticators of mucositis occurring in the healthy oral tissues of H&N cancer patients receiving treatment, and to understand the cytokines balance mechanism of action.

Assuming there is a correlation between high cytokines levels during inflammation and the severity of radiation induced mucositis, finding these prognostic factors may help us predict during the first part of the treatment the need for PEG, placing it prior to the complications associated with severe mucositis on one hand, and avoiding unnecessary procedures on the other hand. This study may also lead to a new strategy of assessing severity of mucositis by laboratory tests, a tool that can be used as an objective assessment in developing strategies that aim to reduce the mucositis. The understanding of the cytokines balance in this condition can also be translated to the use of anti-cytokine treatment for this condition, similar to other immune related diseases such as RA, Crohn's Disease and MS.

Secondary aims of this study are to measure recently available tumor markers SCC and TPS, and to correlate them with tumor response. Genetic markers will be assessed for extreme alteration in radiation reactions such as severe skin reaction, early and unexpectedly severe mucositis, and on the other hand - lack of response. The blood for these tasks will be collected prospectively, but evaluated at the end of the study.

The study will comprise of at least 14 and up to 35 patients with H&N epithelial cancer.

Patients will be clinically evaluated during the week before treatment, and during the treatment period weekly.

Blood samples will be drown for cytokines prior to treatment, at week 2, 4 and at the end of the treatment. The serum collected will be separated for the following factors:

1. Inflammatory Cytokines: IL-1, IL-6, IL-8, IL-18 and TNF α.
2. Anti inflammatory cytokines: IL-10 and TGF β.
3. Tumor markers: SCC and TPS.
4. Genetic assessment of genes that may be involved in extreme treatment reaction. At each weekly follow up, patients will be assessed for mucositis by physician using the WHO common toxicity criteria, and will answer a mucositis questionnaire (based on the RTOG/EORTC questionnaire). Patient's weight will also be recorded.

Scientific aims

The primary aims:

1. To investigate the relationship between cytokine level and the clinically suggested PEG at the end of the H&N chemo-irradiation.
2. To investigate whether a correlation exists between blood cytokines (inflammatory versus anti-inflammatory cytokines) levels and the severity of radiation induced mucositis in patients receiving chemo-radiotherapy for cancer of the H&N.
3. To investigate whether blood cytokines levels could serve as a simple laboratory tool, to predict the severity of mucositis and dysphagia occurring during H&N chemo-irradiation.

The secondary aims:

1. To study the clinical usefulness of the Tumor Markers SCC and TPS in this setting, namely, to evaluate the correlation between their blood levels and response to therapy.
2. To compare the associated mucositis between two commonly used radiation treatment strategies - IMRT 5 field plan and classic two dimensional plan for the subgroup of patients with advanced glottic and supraglottic cancer.
3. To assess whether cytokine levels during treatment can predict long term treatment related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with H&N epithelial cancer (nasopharynx, oropharynx, oral cavity - tongue, buccal mucosae and palate, larynx and hypopharynx)
* Treated with definitive chemo-radiation treatment and follow up
* Male and female patients will be included, with an age ranging between 18- 85 years

Exclusion Criteria:

* Soldiers, prisoners and pregnant women will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Study Completion 2011-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amichay Meirovitz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Wong PC, Dodd MJ, Miaskowski C, Paul SM, Bank KA, Shiba GH, Facione N. Mucositis pain induced by radiation therapy: prevalence, severity, and use of self-care behaviors. J Pain Symptom Manage. 2006 Jul;32(1):27-37. doi: 10.1016/j.jpainsymman.2005.12.020. PMID 16824982
- [Background] Nagler RM, Barak V, Nagler A. Short-term systemic effects of head and neck irradiation. Anticancer Res. 2000 May-Jun;20(3A):1865-70. PMID 10928120
- [Background] Scully C, Epstein J, Sonis S. Oral mucositis: a challenging complication of radiotherapy, chemotherapy, and radiochemotherapy: part 1, pathogenesis and prophylaxis of mucositis. Head Neck. 2003 Dec;25(12):1057-70. doi: 10.1002/hed.10318. PMID 14648865
- [Background] Wood K. Audit of nutritional guidelines for head and neck cancer patients undergoing radiotherapy. J Hum Nutr Diet. 2005 Oct;18(5):343-51. doi: 10.1111/j.1365-277X.2005.00632.x. PMID 16150130
- [Background] Whicher JT, Evans SW. Cytokines in disease. Clin Chem. 1990 Jul;36(7):1269-81. PMID 2197032
- [Background] Peterman A, Cella D, Glandon G, Dobrez D, Yount S. Mucositis in head and neck cancer: economic and quality-of-life outcomes. J Natl Cancer Inst Monogr. 2001;(29):45-51. doi: 10.1093/oxfordjournals.jncimonographs.a003440. PMID 11694566
- [Background] Barak V, Kalickman I, Nisman B, Farbstein H, Fridlender ZG, Baider L, Kaplan A, Stephanos S, Peretz T. Changes in cytokine production of breast cancer patients treated with interferons. Cytokine. 1998 Dec;10(12):977-83. doi: 10.1006/cyto.1998.0378. PMID 10049522